CLINICAL TRIAL: NCT06776250
Title: A Phase II Study Evaluating the Safety, Efficacy, and Intracranial Activity of Tarlatamab in Recurrent/Refractory Gliomas With IDH Mutation (TARGID)
Brief Title: Study of How Safe and Effective Tarlatamab is in Brain Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGID; CAPCR 24-5801 (Other: University Health Network)
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Astrocytic Tumor; Oligodendroglial Tumor
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients whose disease is amendable for resection will be treated with up to 3 cycles of tarlatamab prior to surgical resection. These patients can resume tarlatamab treatment post-operatively until disease progression at the discretion of the investigator. Up to 10 patients may be enrolled to Cohort 1.
  Interventions: Drug: Tarlatamab
- Cohort 2 (Experimental): Patients with progressive/refractory disease are eligible to receive tarlatamab at every 2 weeks 10 mg dosing in 28 day cycles until documented disease progression, intolerable toxicity or consent withdrawal. Up to 34 patients may be enrolled to Cohort 2.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab is a BiTE molecule designed to direct T effector cells toward DLL3-expressing cells.

SUMMARY:
This is a phase 2 study to assess how useful study drug tarlatamab is for the treatment of patients with recurrent/refractory oligodendroglioma or astrocytoma with a mutation in the IDH gene.

DETAILED DESCRIPTION:
There will be 2 cohorts in the study.

* Cohort 1, patients whose disease is amendable for resection will be treated with up to 3 cycles of tarlatamab prior to surgical resection. These patients can resume tarlatamab treatment post-operatively until disease progression at the discretion of the investigator. Up to 10 patients may be enrolled to Cohort 1.
* Cohort 2, patients with progressive/refractory disease are eligible to receive tarlatamab at Q2W 10 mg dosing in 28 day cycles until documented disease progression, intolerable toxicity or consent withdrawal. The Simon's 2 stage design will be used. In stage 1, 13 patients will be enrolled. Based on an interim analysis of efficacy, stage 2 will aim to enroll an additional 21 patients for a total of 34 patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Must be 18 years of age or older.
* Body weight > 40 kg.
* Patients must have histologically or cytologically confirmed diffuse astrocytic or oligodendroglial tumors by World Health Organization 2016 classification which are IDH mutant.
* Patients could have received up to 2 regimens of systemic therapy after relapse.
* For Cohort 1: Patient must be clinically deemed resectable and a resection is clinically indicated.
* For Cohort 2: Patient must be unresectable or a resection is not clinically indicated at the time of enrollment.
* Patients must have normal organ and bone marrow function measured within 14 days prior to administration of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have a life expectancy ≥ 12 weeks.
* Patients of childbearing potential must have a negative serum pregnancy test within 28 days prior to start of therapy and Day 1 prior to start of therapy.
* All participants must agree to use 2 acceptable methods to prevent pregnancy for study required duration.
* Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* All patients in Cohort 1 and Cohort 2 are required to submit archival tissue. In addition,
* Patients in Cohort 1 must be willing to provide fresh tumor samples at the time of clinically indicated surgical resection/debulking, or willing to undergo post-treatment tumor biopsy.
* Patients in Cohort 2 must be willing to provide tumor samples should they require surgical resection/debulking or undergo clinically indicated tumor biopsy after enrollment in trial.
* Patients in Cohort 2 must have measurable and progressive disease documented within 28 days of start of study treatment
* Patients must be asymptomatic and meet the following criteria:
* At least 28 days after the most recent CNS treatment, clinically stable.
* At least 14 days on stable doses of corticosteroids and/or anti-seizure medications.

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (non-intervention) clinical study or the follow-up period of an interventional study.
* Receipt of any conventional or investigational anticancer therapy within 28 days prior to the first dose of tarlatamab.
* Any previous treatment with tarlatamab.
* Other malignancy within the last 5 years with exceptions.
* Patients receiving any systemic chemotherapy or radiotherapy within 28 days prior to study treatment.
* Unresolved toxicity from prior anti-tumor therapy or prior surgery.
* Major surgery within 28 days of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* History of arterial thrombosis within 12 months of first dose of tarlatamab.
* Patients who are pregnant, lactating, or intend to become pregnant during their participation in this study.
* Patients with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of tarlatamab.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV), or those who have had a solid organ transplant or allogeneic transplant.
* History of hypophysitis or pituitary dysfunction.
* Exclusion of hepatitis infection based on the following results and/or criteria (within 3 months prior to the first dose of tarlatamab):
* Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B).
* Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B.
* Positive hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C.
* Whole blood transfusions within 120 days prior to enrollment to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to treatment).
* Current or prior use of immunosuppressive medications within 14 days before the 1st dose of tarlatamab. Patients receiving systemic corticosteroids must have been on a stable dose of corticosteroids for at least 14 days prior to the 1st dose of tarlatamab.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, celiac disease, and Wegner syndrome) within the last 2 years. Patients with vitiligo, alopecia, Grave's disease, hypothyroidism stable on hormone replacement, or psoriasis not requiring systemic treatment (within the past 3 years) are not excluded.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational products or interpretation of patient safety or study results.
* Receipt of live attenuated vaccines within 30 days prior to the 1st dose of tarlatamab, during the study and for 30 days after the last dose of tarlatamab. Examples include, but are not limited to, vaccines for measles, mumps, and rubella, live attenuated influenza vaccine (nasal), chicken pox vaccine, oral polio vaccine, rotavirus vaccine, yellow fever vaccine, BCG vaccine, typhoid vaccine and typhus vaccine.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice).
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to tarlatamab.
* Patients unable to remain within one hour of study site for additional 48 hours after hospitalization on cycle 1 day 1 and cycle 1 day 8.
* Patients unable to remain within one hour of any hospital for 72 hours after infusion of tarlatamab on cycle 1 day 1 and cycle 1 day 8.
* Patients unable to identify home companion who will cohabitate with subject for 72 hours after infusion of tarlatamab on cycle 1 day 1 and cycle 1 day 8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
Percent change in CD8+ T cell infiltrate | 3 years

SECONDARY OUTCOMES:
Percent change in CD3/CD45RA/RO T cells | 3 years
Percent change in T cell subsets | 3 years
Percentage change in M1 vs M2 macrophage populations | 3 years
Tumour concentrations of tarlatamab | 3 years
Serum concentrations of tarlatamab | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, MD, Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No